CLINICAL TRIAL: NCT02405832
Title: Zinc Lozenges and Their Effect on Postoperative Sore Throat Syndrome: A Randomized, Double-blinded, Placebo-controlled Prospective Study
Brief Title: Zinc Lozenges and Their Effect on Postoperative Sore Throat Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Lydia Grondin, Associate Professor of Anesthesiology and Attending Anesthesiologist, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CHRMS 14-206
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Sore Throat; Post-Operative Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc - active arm (Experimental): Oral administration of a 40 mg elemental zinc (in the form of zinc sulfate) lozenge, with sweetener and citrus flavor
  Interventions: Dietary Supplement: Zinc
- Placebo (Placebo Comparator): Placebo lozenge, with sweetener and citrus flavor, administered orally
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc — Oral administration of a 40 mg elemental zinc (in the form of zinc sulfate) lozenge, with sweetener and citrus flavor
  Arms: Zinc - active arm
Dietary Supplement: Placebo — Placebo lozenge, with sweetener and citrus flavor, administered orally
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the effect of preoperative administration of oral zinc lozenges on the incidence of postoperative sore throat syndrome.

When patients undergo surgery with general anesthesia, they require ventilation of their lungs with the help of a flexible tube (called an endotracheal tube) that is placed through the mouth, passing the vocal cords, and into the windpipe (trachea). This tube helps oxygenate the patient, delivers anesthetic gas to the lungs, and keeps the airways open to prevent asphyxiation. The procedure is invasive and uncomfortable, and one of the most common consequences is a sore and inflamed throat after the tube is taken out. This is termed postoperative sore throat (POST). Though the intensity and severity of sore throat varies from person to person, the reported incidence is as high as 90% of patients undergoing general anesthesia.

Zinc therapy has been shown in multiple studies to reduce the severity and duration of cold symptoms, and also to up-regulate the immune system. Recent studies have shown that zinc can act as an anti-inflammatory agent and can maintain the integrity of skin and mucosal membranes (which cover the inside of the mouth and throat). The aim of this study is to evaluate the effects of giving zinc lozenges before tube placement on postoperative sore throat.

After written informed consent is received in pre-op, a sealed and coded envelope with either the zinc lozenge or the placebo lozenge will be given to the patient to be administered orally, with the instruction to dissolve the lozenge by sucking on it 30 minutes prior to surgery. Upon completion of surgery and emergence from general anesthesia, the patient will be extubated and transferred to the post-anesthesia care unit (PACU). Once in the PACU, the patient will be assessed regarding the incidence and severity of POST by the study investigator using a standardized scale. The severity of POST will be graded on a 4-point scale ranging from 0 to 3; 0 being no sore throat, 1 being mild discomfort (complains only upon questioning), 2 being moderate sore throat (complains on his/her own), and 3 being severe sore throat (change in voice, hoarseness, and throat pain). This evaluation will be performed at 30 minutes, 2 hours, 4 hours, and 24 hours post-surgery, with the assessment at 4 hours being the primary outcome of the study.

DETAILED DESCRIPTION:
The overall purpose of this study is to investigate the effects of preoperative administration of oral zinc lozenges on postoperative sore throat syndrome which consists of pain, dysphagia, and in extreme cases hoarseness. It is associated with coughing (which may increase surgical related pain) and difficulty with oral intake. The study will look at the changes in incidence and severity of POST in the immediate postoperative period.

Postoperative sore throat (POST) syndrome is a very common complication of endotracheal intubation Prior to earlier studies larger endotracheal tubes were utilized for providing general anesthesia. The incidence of POST at that time was 48%, with smaller tubes the incidence decreased to 22%. It is now standard of care to utilize endotracheal tubes based on size and gender of the patient. In subsequent studies to further reduce the incidence of POST, the rate of sore throat in the control groups have been between 17-90%. The cause of POST is related to direct local tissue trauma leading to inflammation of the pharyngeal mucosa and possibly the drying effect of non-humidified gases across the mucous membranes. Although there have been multiple treatments recommended for POST, none of them have been exactly effective, and the symptoms usually ameliorate within 72 hr without treatment. Even though this is the case, it is still recommended to take preventive measures for POST. The presence of POST after surgery is a patient satisfaction issue and has also been associated with a longer stay in in the post anesthesia recovery unit(Higgins et al). Both pharmacologic and non-pharmacologic measures have been recommended in past studies. Nonpharmacological methods for attenuating POST have included using smaller-sized endotracheal tubes, lubricating the endotracheal tube with water-soluble jelly, careful airway instrumentation, and minimizing cuff pressure. Pharmacologic measures have included gargles with lidocaine, aspirin, or ketamine preoperatively, inhalation of beclomethasone or fluticasone propionate, and recently the use of licorice gargle or magnesium lozenges 30 min preoperatively (Ruetzler, Borazan H).

Zinc has been utilized for many years as a topical agent to promote epithelial health and recovery after injury. Several studies have evaluated the effect of zinc on wound healing and epithelial tissue health. These studies have shown that supplementation with zinc sulfate causes rapid recovery of leg and gastric ulcers (Worthington et al). It seems zinc not only increases re-epithelialization, but it also decreases bacterial activity and causes rapid wound healing (Arbabi-kalati et al). Zinc has also been shown to be an immunomodulatory agent that monitors and modifies the immune system and T-lymphocytes. Decreases in zinc serum levels lead to lymphopenia and declines in cellular and humoral immunity. The effect of oral zinc sulfate has also been utilized for treatment of oral wounds by oral surgeons; moreover, research has shown zinc supplementation assists with the recovery of mucosal wounds and treatment of tongue ulcers (Worthington et al). A recent study by Arbabi-kalati, showed that high dose oral zinc sulfate (220 mg TID) decreased the intensity of mucositis, xerostomia, and pain in individuals undergoing chemotherapy or radiotherapy treatments. The mechanism by which zinc improves tissue health was investigated by Sharir et al. and in a model of epithelial injury showed that topical zinc directly activates receptors that promote epithelial repair.

Keeping the above studies in mind, the investigators built this study using the protocols devised by Borazan H, in which they evaluated the efficacy of magnesium lozenges on POST. There are currently no known studies that look at the efficacy of zinc in the prevention of POST. The investigators will use custom compounded lozenges from a local pharmacy with 40 mg of elemental zinc (equivalent to 174 mg of zinc sulfate) per lozenge, which is the tolerable upper intake level for zinc in adults as defined by the US department of Food and Nutrition Board.

The possible knowledge gained from this study for POST syndrome can be extended to people undergoing surgeries requiring endotracheal intubation in the future.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 and older
* American Society of Anesthesiologists physical status classification system I and II (healthy patient or patient with mild systemic disease)
* Patient coming for elective surgery (except head and neck) requiring general anesthesia
* Patients staying for at least 24 hours postoperatively
* Patients provide informed consent
* Patients presenting for surgery >1 hour in length and <6 hours.

Exclusion Criteria:

* History of preoperative sore throat, common colds, upper respiratory infections, immune deficiencies
* Chronic smokers
* Patients with Mallampati airway grade of more than 2
* Patients requiring more than one attempt for intubation or traumatic intubations
* Patients requiring laryngeal mask Airway (LMA) placement
* Patients allergic to zinc
* Patients requiring quinolones or tetracycline antibiotics pre- or intraoperatively
* Patients undergoing head and neck surgeries
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2015-04-04 (Actual); Study Completion 2015-04-04 (Actual)

PRIMARY OUTCOMES:
Severity of Post-Operative Sore Throat | 4 hours
  The severity of POST will be graded on a 4-point scale ranging from 0 to 3; 0 being no sore throat, 1 being mild discomfort (complains only upon questioning), 2 being moderate sore throat (complains on his/her own), and 3 being severe sore throat (change in voice, hoarseness, and throat pain).

SECONDARY OUTCOMES:
Severity of Post-Operative Sore Throat at 30 minutes | 30 minutes
  The severity of Post-Operative Sore Throat was graded on a 4-point scale ranging from 0 to 3:
  0 = no sore throat
  1. = mild discomfort (patient complains only upon questioning)
  2. = moderate sore throat (patient complains on their own)
  3. = severe sore throat (change in voice, hoarseness, and throat pain).
Severity of Post-Operative Sore Throat at 2 hours | 2 hours
  The severity of Post-Operative Sore Throat was graded on a 4-point scale ranging from 0 to 3:
  0 = no sore throat
  1. = mild discomfort (patient complains only upon questioning)
  2. = moderate sore throat (patient complains on their own)
  3. = severe sore throat (change in voice, hoarseness, and throat pain).
Severity of Post-Operative Sore Throat at 24 hours | 24 hours
  The severity of Post-Operative Sore Throat was graded on a 4-point scale ranging from 0 to 3:
  0 = no sore throat
  1. = mild discomfort (patient complains only upon questioning)
  2. = moderate sore throat (patient complains on their own)
  3. = severe sore throat (change in voice, hoarseness, and throat pain).

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Grondin, M.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbabi-kalati F, Arbabi-kalati F, Deghatipour M, Ansari Moghadam A. Evaluation of the efficacy of zinc sulfate in the prevention of chemotherapy-induced mucositis: a double-blind randomized clinical trial. Arch Iran Med. 2012 Jul;15(7):413-7. PMID 22724877
- [Background] Borazan H, Kececioglu A, Okesli S, Otelcioglu S. Oral magnesium lozenge reduces postoperative sore throat: a randomized, prospective, placebo-controlled study. Anesthesiology. 2012 Sep;117(3):512-8. doi: 10.1097/ALN.0b013e3182639d5f. PMID 22797283
- [Background] Higgins PP, Chung F, Mezei G. Postoperative sore throat after ambulatory surgery. Br J Anaesth. 2002 Apr;88(4):582-4. doi: 10.1093/bja/88.4.582. PMID 12066737
- [Background] Ruetzler K, Fleck M, Nabecker S, Pinter K, Landskron G, Lassnigg A, You J, Sessler DI. A randomized, double-blind comparison of licorice versus sugar-water gargle for prevention of postoperative sore throat and postextubation coughing. Anesth Analg. 2013 Sep;117(3):614-621. doi: 10.1213/ANE.0b013e318299a650. Epub 2013 Aug 6. PMID 23921656
- [Background] Sharir H, Zinger A, Nevo A, Sekler I, Hershfinkel M. Zinc released from injured cells is acting via the Zn2+-sensing receptor, ZnR, to trigger signaling leading to epithelial repair. J Biol Chem. 2010 Aug 20;285(34):26097-106. doi: 10.1074/jbc.M110.107490. Epub 2010 Jun 3. PMID 20522546
- [Background] Worthington HV, Clarkson JE, Bryan G, Furness S, Glenny AM, Littlewood A, McCabe MG, Meyer S, Khalid T. Interventions for preventing oral mucositis for patients with cancer receiving treatment. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD000978. doi: 10.1002/14651858.CD000978.pub3. PMID 21154347
- [Derived] Farhang B, Grondin L. The Effect of Zinc Lozenge on Postoperative Sore Throat: A Prospective Randomized, Double-Blinded, Placebo-Controlled Study. Anesth Analg. 2018 Jan;126(1):78-83. doi: 10.1213/ANE.0000000000002494. PMID 28953493